CLINICAL TRIAL: NCT02736786
Title: A Study of Mucosal Sparing Proton Beam Therapy (PBT) in Resected Oropharyngeal Tumors
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Samir Patel, Assistant Professor of Radiation Oncology, Mayo Clinic
Other Study IDs: 16-000040
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Oropharyngeal Tumor
Keywords: proton
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is an observational study evaluating the clinical outcomes of mucosal sparing proton beam therapy (PBT) after resection of favorable risk oropharyngeal cancer patients. Subjects will be screened at outpatient clinic visit appointments and interested qualified subjects will be consented and offered participation in this study. Once consent has been obtained baseline adverse event and Quality of Life (QOL) data will be collected and subjects will undergo adjuvant PBT and follow-up at 3 months, 12 months, and 24 months. No study-specific visits or evaluations will be required. Patients will be evaluated according to the physician's standard practice and discretion. Patient data will be drawn from the patients' medical records and reported by means of a web-based electronic data collection (EDC) system. Patients will be considered "on study" until 24 months of observation has occurred, withdrawal of consent, lost to follow-up, or study closure.

ELIGIBILITY:
Inclusion Criteria:

* Resection of oropharyngeal tumor by transoral surgery using frozen section margin analysis resulting in a negative margin resection
* No extensive perineural invasion after review by head and neck pathologist
* No lymphovascular invasion after review by head and neck pathologist
* Pathologic stage T1-2 N1-3 M0 disease

Exclusion Criteria:

* T3 or T4 primary stage disease
* Prior radiation therapy to the head and neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Oropharyngeal cancer resected using transoral surgery with positive lymphadenopathy requiring adjuvant radiation therapy.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Local Control Rate in Patients Treated with Proton Beam Therapy after Resection Using Transoral Surgery | 24 months
  Local control rate will be assessed by standard of care head and neck clinical examination during routine followup visits

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials